CLINICAL TRIAL: NCT02733133
Title: A Single-Dose, Single Period, Phase II Pharmacokinetic Study To Examine Testagen™ TDS®-Testosterone For Its Potential To Be Inadvertently Transferred By Skin Contact After Dosing In Healthy Adult Subjects
Brief Title: Product Transference Study of Testagen™ TDS®-Testosterone
Acronym: TRANSFERENCE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Transdermal Delivery Solutions Corp (Industry)
Collaborators: Advanced Therapies Centre, The London Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PARC-Testosterone-T1/09/13; 2013-001767-23 (EudraCT Number); IRAS project ID: 146877 (Other: London - West London & GTAC Research Ethics Committee)
Record Dates: First submitted 2016-03-10; First posted 2016-04-11 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-01

CONDITIONS: Hypogonadotropism
Keywords: Testosterone; AndroGel; Transference; Women; Children
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Uncovered (Experimental): Half of the male partners in each cohort will apply the Testagen® TDS Testosterone 5% HypoSpray® and cover the area before engaging in contact with the female partner.
  Interventions: Drug: Testagen® TDS Testosterone 5% HypoSpray®
- Covered (Experimental): Half of the male partners in each cohort will apply the Testagen® TDS Testosterone 5% HypoSpray® and will not cover the area before engaging in contact with the female partner.
  Interventions: Drug: Testagen® TDS Testosterone 5% HypoSpray®

INTERVENTIONS:
Drug: Testagen® TDS Testosterone 5% HypoSpray® — Topically applied Testosterone Hormone Replacement Lotion

SUMMARY:
This study will assess the potential of Testagen® TDS-Testosterone to enable transfer of Testosterone to females coming in contact with skin to which Testagen® TDS-Testosterone has been applied and the potential of product to raise serum androgen levels in those women.

DETAILED DESCRIPTION:
48 Couples will be added to the protocol and a single dose applied by the male member of the couple. The female member of the couple will have undergone a baseline pharmacokinetic monitoring of her endogenous levels of Testosterone. At precise intervals by cohort on the day of the trial, the male will expose the skin onto which the trial materials were applied to the skin of his partner and she will then undergo another 24-hour multiple sample monitoring of her levels of testosterone.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Volunteers
2. Subject Couples, between 18 and 80 years of age, inclusive.
3. The subject couple is willing and able to read, understand the Subject Information Sheets and provide written informed consent.
4. The subject has a body mass index (BMI) within 18-30 kg/m2.
5. The subject is in otherwise good health as determined by medical history and physical examination.
6. Female subjects must be practicing an acceptable method of birth control. Acceptable methods of birth control include hormonal contraceptives. If practicing an acceptable method of birth control, a negative urine pregnancy test result has been obtained on each Treatment Day.
7. The subject is a non-smoker.
8. The female subject must agree to comply with the placement of an indwelling catheter on two separate occasions and the drawing of blood samples for the pharmacokinetic assessments.
9. The subject couple is willing and able to comply with all testing and requirements defined in the protocol.
10. The subject couple is willing and able to return to the study site for all visits.

Exclusion Criteria:

1. The subject has any relevant deviations from normal in physical examination, electrocardiogram (ECG), or clinical laboratory tests, as evaluated by the investigator, particularly an elevated PSA reading or positive pregnancy test.
2. The subject has had a clinically significant illness within 30 days preceding entry into this study.
3. The subject has a history of significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, or metabolic disease.
4. The subject has a known allergy or history of hypersensitivity to Testosterone or similar compounds.
5. The subject has used any prescription medication within 14 days or over-the-counter (OTC) medication or alcohol within 48 hours of dosing or intends to use any prescription or OTC medication during the study that may interfere with the evaluation of study medication (excluding oral contraceptives).
6. The subject has donated or lost a significant volume of blood (>450mL) within four (4) weeks of the study, and their haemoglobin concentration and haematocrit have not returned to within 5% of normal.
7. The subject has a history of substance abuse or a current positive urine drug screen.
8. Alcohol consumption greater than community norms (i.e. more than 21 standard drinks per week for males, and 14 for females).
9. Subjects who have received an investigational drug or have used an investigational device in the 30 days prior to study entry.
10. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2016-11; Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Transference of Topical Testosterone from Dosed Males to Female Partners As Measured by net change from Baseline of Serum Testosterone in nG/dL expressed as Maximum Serum Concentration or Cmax. | 30 minutes to 24 hours post dose
  Determination of whether testosterone from the Testagen® preparation is transferable from the skin of the patient to his partner and therefore detectable in the blood of female partner and if so, how much as measured by ELISA method as applied to blood samples and computed for Concentration Max (Cmax) for 24 hours post dose measured in ng/dL Testosterone as determined by ELISA method.

SECONDARY OUTCOMES:
Transference of Topical Testosterone from Dosed Males to Female Partners As Measured by net change from Baseline of Serum Testosterone in nG/dL expressed as Area Under Curve or AUC. | 30 minutes to 24 hours post dose
  Determination of whether testosterone from the Testagen® preparation is transferable from the skin of the patient to his partner and therefore detectable in the blood of female partner and if so, how much as measured by ELISA method as applied to blood samples and computed for Area Under the Curve (AUC) for 24 hours post dose measured in ng/dL Testosterone as determined by ELISA method.

OTHER OUTCOMES:
Transference of Topical Testosterone from Dosed Males with application area covered to Female Partners As Measured by net change from Baseline of Serum Testosterone in nG/dL expressed as Maximum Serum Concentration or Cmax | 30 minutes to 24 hours post dose
  Determination of whether testosterone from the Testagen® preparation is transferable from the skin of the patient with application area covered to his partner and therefore detectable in the blood of female partner and if so, how much as measured by ELISA method as applied to blood samples and computed for Concentration Max (Cmax) and Area Under the Curve (AUC) for 24 hours post dose measured in ng/dL Testosterone as determined by ELISA method.
Transference of Topical Testosterone from Dosed Males with application area covered to Female Partners As Measured by net change from Baseline of Serum Testosterone in nG/dL expressed as Area Under the Curve or AUC | 30 minutes to 24 hours post dose
  Determination of whether testosterone from the Testagen® preparation is transferable from the skin of the patient and therefore detectable in the blood of the female partner with application area covered to his partner and if so, how much as measured by ELISA method as applied to blood samples and computed Area Under the Curve (AUC) for 24 hours post dose measured in ng/dL Testosterone as determined by ELISA method.

CONTACTS AND LOCATIONS:
Overall Officials: Shern L. Chew, M.D., Ph.D., Principal Investigator — Consultant Physician and Professor of Endocrine Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Chik Z, Johnston A, Tucker AT, Chew SL, Michaels L, Alam CA. Pharmacokinetics of a new testosterone transdermal delivery system, TDStestosterone in healthy males. Br J Clin Pharmacol. 2006 Mar;61(3):2759. — https://www.ncbi.nlm.nih.gov/pubmed/16487220?dopt=Abstract